CLINICAL TRIAL: NCT01469260
Title: Effective Pedometer Use to Prevent Excessive Gestational Weight Gain in Overweight/Obese Women
Brief Title: Pedometer Use to Prevent Excessive Pregnancy Weight Gain in Overweight Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: resources
Sponsor: Stanford University (Other)
Collaborators: Lucile Packard Children's Hospital (Other)
Responsible Party: Principal Investigator, Susan D Crowe, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22651
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Overweight; Obesity; Pregnancy
Keywords: Overweight; Obesity; Pregnancy; Weight gain; Pedometer; Exercise
MeSH Terms: conditions — Overweight; Obesity; Weight Gain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine care (No Intervention): ACOG Exercise in Pregnancy pamphlet
- Pedometer (Experimental): ACOG Exercise in Pregnancy pamphlet, pedometer use, ultimate goal of 10,000 steps per day
  Interventions: Other: Pedometer

INTERVENTIONS:
Other: Pedometer — Pedometer provided, counseling on pedometer use and step recommendations of 10,000 steps per day, handouts given every 4 weeks to encourage exercise
  Arms: Pedometer

SUMMARY:
The purpose of this study is to evaluate pedometer use by overweight women during pregnancy. The study will show if a pedometer will help women to limit weight gain during pregnancy. It will also show if it there are other benefits such as decreased diabetes, decreased high blood pressure, decreased rates of cesarean section, and decreased complications for the baby.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Pregnant
* Less than 16 weeks gestation
* Body mass index 25 or greater at first prenatal visit

Exclusion Criteria:

* History of spontaneous preterm delivery between 20-32 weeks gestation
* Medical contraindication to exercise or walking during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
Excessive gestational weight gain | At delivery
  Gestational weight gain greater than Institute of Medicine recommendations

SECONDARY OUTCOMES:
Postpartum weight | 6 weeks postpartum
Weight at 1 year postpartum | 1 year postpartum
Gestational diabetes | During pregnancy
Hemoglobin A1c | 24-28 weeks gestation
Infant birth weight | At delivery
Mode of delivery | At delivery
Hypertensive disorders of pregnancy | During pregnancy
Neonatal intensive care unit admission or neonatal complications | Up to 1 week after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Susan Crowe, MD, Principal Investigator — Stanford University; Joyce Sung, MD, Study Chair — Stanford University
Locations (1):
- Lucile Packard Children's Hospital Obstetrics Clinic, Palo Alto, California, United States